CLINICAL TRIAL: NCT04038424
Title: The Effect of Art Therapy on Cognitive Ability, Arm Activity and Mental Health Status in Patients With Stroke
Brief Title: The Effect of Art Therapy on Patients With Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Naglaa Fathy Afifi Youssef, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-44
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke and Hemorrhagic Stroke
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke | interventions — Art Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The intervention group (n = 30) will receive Routine Hospital Management (RHM), conventional rehabilitation activity and AT (painting, coloring, listening to music and Hand Therapy Ball Exercises). Overall 9 sessions over a period of three weeks will be performed and each session will take around 30 min.
  Interventions: Other: Art therapy
- Control group (No Intervention): The control group (n = 30) will receive only the Routine Hospital Management (RHM) and the department conventional rehabilitation activity.

INTERVENTIONS:
Other: Art therapy — Art therapy including coloring, painting and listening to music
  Other Names: Hand Therapy Ball Exercises
  Arms: Study group

SUMMARY:
Stroke can affect the physical, emotional and social aspects of the patient and their family members. It is the main cause of complex disability, with a high number of people living with its effects. Stroke can result in impairments in motor function, language, cognition, sensory processing, cognition, and emotional disturbances, which can affect the performance of functional activities and mental health status. Getting patients involved in art therapy (AT) class has shown to alleviate stress and promote a sense of wellbeing, which can aid their recovery and rehabilitation. The benefits of art therapy for people living with different health conditions worldwide have been reported, however, its effect on Egyptian patients with stroke has been neglected.

DETAILED DESCRIPTION:
Art therapy refers to a group of techniques including painting, drawing and listening to music. The participants will receive the program on three steps (early step, middle step, and late step). These steps aim to train the participants on the AT from simple to complex and motivate them to engage in the AT program.Therefore, this study aims to investigate the effect of art therapy on cognitive ability, arm activity and mental health status of patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* able to sit upright, supported or unsupported,
* oriented to time and place by using the adapted Arabic Memory Screening Test,
* able to perform at least two of the following skills: drinking from a cup, eating with a spoon and taking money from a purse by the affected arm, and
* will stay in the stroke unit to at least 4 days (for receiving three sessions out of all sessions) before discharge,

Exclusion Criteria:

* diagnosis of transient ischemic attack or brain stem stroke;
* unconscious;
* unable to provide informed consent;
* hemodynamical unstable medical conditions, including fever;
* serious infectious diseases, for example, viral hepatitis or HIV; and/or
* severe dementia or uncontrolled psychiatric problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The Montreal Cognitive Assessment (MOCA) | 3 weeks
  The Montreal Cognitive Assessment is a 16-item screening assessment for mild cognitive impairment. It is widely used in stroke survivors and assesses performance attention, concentration, executive functions, memory, language, visual-constructional skills, conceptual thinking, calculations and orientation. The maximum score is 30 and scores of under 26 indicate cognitive impairment.
The Hospital Anxiety and Depression Scale (HADS) | 3 weeks
  This measurement consists of two subscales: Anxiety subscale (HADS-A) and a depression subscale (HADS-D) with 14 intermingled items. Each item is rated on a four-point scale of 0-3, giving maximum scores of 21 for anxiety and depression respectively. Scores of 11 or more on either subscale are considered as significant 'case' of psychological comorbidity, a score of 8-10 as borderline while a score of 7 or below is considered as normal.
The Arm Activity (ArmA) Measure | 3 weeks
  The ArmA measure is a patient and/or career-reported 20-item measure of difficulty in passive and active hemiparetic arm function. It consists of a seven-item passive function subscale, and 13-item active function subscale. Using a Likert scoring system between zero (no difficulty) and four (unable to do task). The passive function subscale scores range from zero (high function) to 28 and the active function subscale scores range from zero (high function) to 52.

SECONDARY OUTCOMES:
The Roger's Happy Sad face | pre and post each session/3 weeks
  This Roger's scale will be used to assess mood, anxiety, and pain. The score ranges from 0-4, with 0 ''no symptoms'', and 4 ''worst possible symptoms''.
Self-efficacy and satisfaction for Art | 3 weeks
  To assess self-efficacy and perceived difficulty for art expression we will ask two single item questions. a four-point visual analogue scale with one as least confident/difficult and four as most confident/difficult. Additional question will be asked to rate the participant satisfaction with the intervention as a supportive method during their treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of stroke and cerebral vascular disease treatment, Cairo, Egypt